CLINICAL TRIAL: NCT04324203
Title: The Effectiveness of 3DVR Horticultural Therapy on Older Adults' Physical and Mental Health
Brief Title: The Effectiveness of 3DVR Horticultural Therapy on Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201710HM006
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Physical Health; Mental Health
Keywords: Horticultural therapy; 3D VR; Older adults; long-term care facility; mental health
MeSH Terms: conditions — Psychological Well-Being | interventions — Horticultural Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Three-dimensional Virtual Reality and Horticultural Therapy
  Interventions: Other: Three-dimensional Virtual Reality and Horticultural Therapy
- Control group (No Intervention): No intervention

INTERVENTIONS:
Other: Three-dimensional Virtual Reality and Horticultural Therapy — VR is a realistic, three-dimensional, and virtual environment formed by a combination of computer software and hardware
  Arms: Experimental group

SUMMARY:
This study intends to develop a 3DVR-based horticultural therapy intervention to explore the health effectiveness among older adults

DETAILED DESCRIPTION:
Background: Institutionalized older adults have limited ability to engage in horticultural activities that can promote their physical and mental health.

Objective: This study explored the effects of a combination of three-dimensional (3D) virtual reality (VR) and horticultural therapy (HT) on institutionalized older adults' physical and mental health.

Methods: The study applied a quasi-experimental design. A total of 106 older adults from two long-term care facilities were recruited and assigned to the experimental (n = 59) or control (n = 47) group. The experimental participants received a nine-week intervention. Both groups completed three assessments: at baseline, after the intervention, and two months later. The outcome variables included health status, meaning in life, perceived mattering, loneliness, and depression.

ELIGIBILITY:
Inclusion Criteria:

* over 65 years old.
* being a long-term resident of the selected LTCF
* possessing the ability to understand verbal meanings
* being able to freely operate a joystick.

Exclusion Criteria:

* a history of severe psychiatric conditions, dementia, significant visual or hearing impairment, and/or current severe illnesses such as stroke or Parkinson's disease.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Health Status | Two months
  To assess the health status of the elderly participants, we used the Chinese Health Scale (CHQ-12). This scale consists of 12 Likert-type items that are scored from 3 (not at all) to 0 (more than usual). The higher the score, the higher the level of general health.
Meaning in life. | Two months
  The meaning in life questionnaire was adapted from the purpose in life (PIL) survey, and it consists of 9 Likert-type items. Each item is scored on a Likert-type scale from 1-5, with higher scores indicating a higher level of perceived meaning in life.
Perceived mattering | Two months
  Perceived mattering was adapted from the General mattering Scale (GMS), and consisted of five items. Each item was scored on a Likert-type scale of 1(not at all) to 4(very much) with higher scores indicating a higher level of perceived mattering.
Loneliness | Two months
  The short-form UCLA Loneliness Scale (ULS-6), which consists of six items, was used to measure loneliness. Each item was reversely scored on a Likert-type scale from 4 (never) to 1 (often), with higher scores indicating a lower level of perceived loneliness.
Depression | Two months
  Using a Chinese version of the short-form of the Geriatric Depression Scale (GDS-15). The total raw score ranged from 0-15, with a higher score indicating a lower level of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Long Guo, Principal Investigator — National Taiwan Normal University
Locations (1):
- National Taiwan Normal University,, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bossen A. The importance of getting back to nature for people with dementia. J Gerontol Nurs. 2010 Feb;36(2):17-22. doi: 10.3928/00989134-20100111-01. Epub 2010 Feb 5. PMID 20128524
- [Background] Cheng TA, Williams P. The design and development of a screening questionnaire (CHQ) for use in community studies of mental disorders in Taiwan. Psychol Med. 1986 May;16(2):415-22. doi: 10.1017/s0033291700009247. PMID 3726013
- [Background] Lee IM, Paffenbarger RS Jr, Hennekens CH. Physical activity, physical fitness and longevity. Aging (Milano). 1997 Feb-Apr;9(1-2):2-11. doi: 10.1007/BF03340123. PMID 9177581
- [Background] Soderback I, Soderstrom M, Schalander E. Horticultural therapy: the 'healing garden'and gardening in rehabilitation measures at Danderyd Hospital Rehabilitation Clinic, Sweden. Pediatr Rehabil. 2004 Oct-Dec;7(4):245-60. doi: 10.1080/13638490410001711416. PMID 15513768
- [Background] Grazuleviciene R, Vencloviene J, Kubilius R, Grizas V, Danileviciute A, Dedele A, Andrusaityte S, Vitkauskiene A, Steponaviciute R, Nieuwenhuijsen MJ. Tracking Restoration of Park and Urban Street Settings in Coronary Artery Disease Patients. Int J Environ Res Public Health. 2016 May 31;13(6):550. doi: 10.3390/ijerph13060550. PMID 27258294
- [Background] Chan HY, Ho RC, Mahendran R, Ng KS, Tam WW, Rawtaer I, Tan CH, Larbi A, Feng L, Sia A, Ng MK, Gan GL, Kua EH. Effects of horticultural therapy on elderly' health: protocol of a randomized controlled trial. BMC Geriatr. 2017 Aug 29;17(1):192. doi: 10.1186/s12877-017-0588-z. PMID 28851276
- [Background] Han AR, Park SA, Ahn BE. Reduced stress and improved physical functional ability in elderly with mental health problems following a horticultural therapy program. Complement Ther Med. 2018 Jun;38:19-23. doi: 10.1016/j.ctim.2018.03.011. Epub 2018 Mar 28. PMID 29857876
- [Background] Yao YF, Chen KM. Effects of horticulture therapy on nursing home older adults in southern Taiwan. Qual Life Res. 2017 Apr;26(4):1007-1014. doi: 10.1007/s11136-016-1425-0. Epub 2016 Oct 1. PMID 27696109
- [Background] Stern C, Konno R. Physical Leisure Activities and their Role in Preventing Dementia: A Systematic Review. JBI Libr Syst Rev. 2009;7(8):260-308. doi: 10.11124/01938924-200907080-00001. PMID 27820066
- [Background] Chen YM, Ji JY. Effects of Horticultural Therapy on Psychosocial Health in Older Nursing Home Residents: A Preliminary Study. J Nurs Res. 2015 Sep;23(3):167-71. doi: 10.1097/jnr.0000000000000063. PMID 25534575
- [Background] Liu Y, Bo L, Sampson S, Roberts S, Zhang G, Wu W. Horticultural therapy for schizophrenia. Cochrane Database Syst Rev. 2014 May 19;2014(5):CD009413. doi: 10.1002/14651858.CD009413.pub2. PMID 24842458
- [Background] Heinrich LM, Gullone E. The clinical significance of loneliness: a literature review. Clin Psychol Rev. 2006 Oct;26(6):695-718. doi: 10.1016/j.cpr.2006.04.002. Epub 2006 Jun 19. PMID 16952717